CLINICAL TRIAL: NCT01029652
Title: A 12 Weeks Randomized, Controlled Core Study of ACZ885 (Canakinumab) on the Treatment and Prevention of Gout Flares in Patients With Frequent Flares for Whom NSAIDs and/or Colchicine Are Contraindicated, Not Tolerated or Ineffective, Including a 12-week Double-blind Extension Study and an Open-label 48 Week Extension Study
Brief Title: Canakinumab in the Treatment of Acute Gout Flares and Prevention of New Flares in Patients Unable to Use Non-steroidal Anti-inflammatory Drugs (NSAIDs) and/or Colchicine Including a 12 Weeks Extension and an Open-label 48 Weeks Extension Study
Acronym: β-RELIEVED
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CACZ885H2356; 2009-015018-23 (EudraCT Number); CACZ885H2356E1 (Other: Novartis); CACZ885H2356E2 (Other: Novartis); NCT01071213 (obsolete NCT alias); NCT01160016 (obsolete NCT alias)
Record Dates: First submitted 2009-12-09; First posted 2009-12-10 (Estimated); Results first posted 2011-11-18 (Estimated); Last update posted 2014-01-30 (Estimated); Status verified 2012-09

CONDITIONS: Acute Gout
Keywords: frequent flares; gout; anti-interleukin-1β monoclonal antibody
MeSH Terms: conditions — Gout | interventions — canakinumab; Triamcinolone Acetonide

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Canakinumab 150 mg (Experimental): Patients received 1 subcutaneous (sc) injection of canakinumab 150 mg and 1 intramuscular (im) injection of placebo to triamcinolone acetonide on Day 1. Patients could receive re-dose of study drug on demand upon occurrence of new flares, but re-dosing could not occur until 14 days had elapsed after previous dose. Patients completing 12 weeks core study were allowed to continue treatment in another 12-week extension for any new gout flare on demand with same treatment as assigned in core study.
  After completing the first extension, patients were offered to enter second extension study, whereby all patients were treated open-label "on demand" with canakinumab 150 mg sc upon new flare for 1 year for a total duration of 18 months following randomization in core study. Patients completing first 12 weeks extension study were allowed to continue to be treated in another single-arm, open-label 48 weeks extension when all patients from both treatment arms received canakinumab on demand
  Interventions: Drug: Canakinumab 150 mg; Drug: Placebo to triamcinolone acetonide
- Triamcinolone acetonide 40 mg (Active Comparator): Patients received 1 intramuscular (im) injection of triamcinolone acetonide 40 mg and 1 subcutaneous (sc) injection of placebo to canakinumab on Day 1. Patients could receive a re-dose of study drug on demand upon the occurrence of new flares, but re-dosing could not occur until 14 days had elapsed after the previous dose. Patients completing the 12 weeks core study were allowed to continue to be treated in another 12 weeks extension study for any new gout flare on demand with the same treatment as assigned in the core study.
  Patients under this arm who agreed to continue to 2nd extension period of 12 months, were switched to canakinumab 150 mg sc for any new gout flare during this period Triamcinolone acetonide was not to be administered in the 48-week session.
  Interventions: Drug: Triamcinolone acetonide 40 mg; Drug: Placebo to canakinumab

INTERVENTIONS:
Drug: Canakinumab 150 mg — Canakinumab 150 mg was supplied in 6 mL glass vials each containing nominally 150 mg canakinumab (plus 20% overfill).
  Arms: Canakinumab 150 mg
Drug: Triamcinolone acetonide 40 mg — Triamcinolone acetonide 40 mg was supplied as a suspension.
  Arms: Triamcinolone acetonide 40 mg
Drug: Placebo to canakinumab — Placebo to canakinumab was supplied in 6 mL glass vials containing placebo powder as a lyophilized cake.
  Arms: Triamcinolone acetonide 40 mg
Drug: Placebo to triamcinolone acetonide — Placebo triamcinolone acetonide was supplied as a lipid emulsion similar in appearance to triamcinolone acetonide.
  Arms: Canakinumab 150 mg

SUMMARY:
The purpose of the 12-week core study was to demonstrate that canakinumab given upon acute gout flares relieves the signs and symptoms and prevents recurrence of gout flares in patients with frequent flares of gout for whom non-steroidal anti-inflammatory drugs (NSAIDs) and/ or colchicine are contraindicated, not tolerated, or ineffective. The efficacy of canakinumab was compared to the corticosteroid triamcinolone acetonide.

The purpose of the first 12-week extension study was to collect additional safety, tolerability and efficacy data in patients who have completed the core study CACZ885H2356.

The purpose of the second 48 week open-label extension study was to collect additional long-term safety and tolerability data in patients who have completed the first extension study CACZ885H2356E1.

DETAILED DESCRIPTION:
Masking:

Core: Double Blind (Subject, Investigator) Extension 1: Double Blind (Subject, Investigator) Extension 2: Open-label, terminated

ELIGIBILITY:
Core Study:

Inclusion criteria:

* Meeting the American College of Rheumatology (ACR) 1977 preliminary criteria for the classification of acute arthritis of primary gout
* Onset of current acute gout flare within 5 days prior to study entry
* Baseline pain intensity ≥ 50 mm on the 0-100 mm visual analog scale (VAS)
* History of ≥ 3 gout flares within the 12 months prior to study entry
* Contraindication, intolerance, or lack of efficacy for non-steroidal anti-inflammatory drugs (NSAIDs) and/or colchicine

Exclusion criteria:

* Rheumatoid arthritis, evidence/suspicion of infectious/septic arthritis, or other acute inflammatory arthritis
* Presence of severe renal function impairment
* Use of specified pain relief medications or biologics ( corticosteroids, narcotics, paracetamol/acetominophen, ibuprofen, colchicine, IL-blocker, and tumor necrosis factor inhibitor) within specified periods prior to study entry
* Live vaccinations within 3 months prior to randomization
* Requirement for administration of antibiotics against latent tuberculosis (TB)
* Refractory heart failure (Stage D)
* Unstable cardiac arrhythmias or unstable symptomatic coronary ischemia
* Any active or recurrent bacterial, fungal, or viral infection

Extension Study 1:

Inclusion Completion of the Core study. A patient was defined as completing the core study if they completed the study up to and including visit 7.

Exclusion

- Continuation in this extension study was considered inappropriate by the treating physician.

Extension Study 2:

Inclusion Completed of the first extension study CACZ885H2356E1. A patient was defined as completing the first extension study if they completed the study up to and including Visit 10).

Exclusion

-Continuation in this extension study was considered inappropriate by the treating physician

Other protocol-defined inclusion-exclusion criteria applied to the core and extension studies.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2009-12; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (47):
- Australia (4):
  - Novartis Investigative Site, Darlinghurst, New South Wales
  - Novartis Investigative Site, Fitzroy, Victoria
  - Novartis Investigative Site, Heidelberg, Victoria
  - Novartis Investigative Site, Daw Park SA
- Novartis Investigative site, Gozée, Belgium
- Canada (3):
  - Novartis Investigative Site, Mount Pearl, Newfoundland and Labrador
  - Novartis Investigative site, St. John's, Newfoundland and Labrador
  - Novartis Investigative site, Hamilton, Ontario
- Colombia (3):
  - Novartis Investigative site, Barranquilla
  - Novartis Investigative site, Bogotá
  - Novartis Investigative site, Bucaramanga
- Estonia (3):
  - Novartis Investigative site, Pärnu
  - Novartis Investigative site, Tallinn
  - Novartis Investigative site, Tartu
- Germany (6):
  - Novartis Investigative Site, Bayreuth
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Löhne
  - Novartis Investigative Site, Magdeburg
  - Novartis Investigative site, Munich
- Novartis Investigative Site, Guatemala City, Guatemala
- Latvia (2):
  - Novartis Investigative Site, Riga
  - Novartis Investigative Site, Valmiera
- Lithuania (5):
  - Novartis Investigative Site, Kaunas
  - Novartis Investigative Site, Kėdainiai
  - Novartis Investigative site, Klaipėda
  - Novartis Investigative Site, Šiauliai
  - Novartis Investigative Site, Vilnius
- Mexico (3):
  - Novartis Investigative site, Culiacán
  - Novartis Investigative site, Guadalajara
  - Novartis Investigative site, Mexicali
- Novartis Investigative site, Oslo, Norway
- Poland (4):
  - Novartis Investigative site, Katowice
  - Novartis Investigative site, Kutno
  - Novartis Investigative site, Lublin
  - Novartis Investigative Site, Wroclaw
- Russia (3):
  - Novartis Investigative site, Moscow
  - Novartis Investigative site, Yaroslavl
  - Novartis Investigative site, Yekaterinburg
- Novartis Investigative site, Singapore, Singapore
- Sweden (2):
  - Novartis Investigative Site, Gothenburg
  - Novartis Investigative site, Stockholm
- Novartis Investigative Site, Lausanne, Switzerland
- Ukraine (4):
  - Novartis Investigative Site, Donetsk
  - Novartis Investigative Site, Kyiv
  - Novartis Investigative Site, Lviv
  - Novartis Investigative Site, Zaporizhzhya

REFERENCES:
- [Derived] Chakraborty A, Van LM, Skerjanec A, Floch D, Klein UR, Krammer G, Sunkara G, Howard D. Pharmacokinetic and pharmacodynamic properties of canakinumab in patients with gouty arthritis. J Clin Pharmacol. 2013 Dec;53(12):1240-51. doi: 10.1002/jcph.162. Epub 2013 Sep 30. PMID 24122883

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two patients randomized to canakinumab did not receive any study medication and were discontinued from the core study on the day of randomization, with the reason for discontinuation listed as Administrative Problems.
Groups:
- Canakinumab 150 mg: Patients received 1 subcutaneous (sc) injection of canakinumab 150 mg and 1 intramuscular (im) injection of placebo to triamcinolone acetonide on Day 1. Patients could receive a re-dose of study drug on demand upon the occurrence of new flares, but re-dosing could not occur until 14 days had elapsed after the previous dose. Patients completing the 12 weeks core study were allowed to continue to be treated in another 12 weeks extension study for any new gout flare on demand with the same treatment as assigned in the core study.
  After completing the first extension study, patients were offered to enter the second extension study, whereby all patients were treated open-label "on demand" with canakinumab 150 mg sc upon new flare for 1 year for a total duration of 18 months following randomization in the core study
- Triamcinolone Acetonide 40 mg: Patients received 1 intramuscular (im) injection of triamcinolone acetonide 40 mg and 1 subcutaneous (sc) injection of placebo to canakinumab on Day 1. Patients could receive a re-dose of study drug on demand upon the occurrence of new flares, but re-dosing could not occur until 14 days had elapsed after the previous dose. Patients completing the 12 weeks core study were allowed to continue to be treated in another 12 weeks extension study for any new gout flare on demand with the same treatment as assigned in the core study.
  Patients under this arm who agreed to continue to 2nd extension period of 12 months, were switched to canakinumab 150 mg sc for any new gout flare during this period. No patient received triamcinolone acetonide in second extension Study .
Period: Core Study (0-12 Weeks)
Arm/Group | Canakinumab 150 mg | Triamcinolone Acetonide 40 mg
Started | 115 | 115
Full Analysis Set (FAS), Safety Set | 113 | 115
Completed | 109 | 105
Not Completed | 6 | 10
Not completed — Unsatisfactory therapeutic effect | 0 | 4
Not completed — Patient Withdrew Consent | 1 | 3
Not completed — Lost to Follow-up | 3 | 1
Not completed — Administrative problems | 2 | 1
Not completed — Death | 0 | 1
Period: Extension Study 1 (12-24 Weeks)
Arm/Group | Canakinumab 150 mg | Triamcinolone Acetonide 40 mg
Started | 90 | 85
Completed | 87 | 80
Not Completed | 3 | 5
Not completed — Unsatisfactory therapeutic effect | 0 | 1
Not completed — Lost to Follow-up | 2 | 3
Not completed — Protocol Deviation | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1
Period: Extension Study 2 (25-72 Weeks)
Arm/Group | Canakinumab 150 mg | Triamcinolone Acetonide 40 mg
Started | 69 | 66
Re-treated With or Switch to Canakinumab | 69 (Includes patients re-treated with canakinumab over 72 weeks study duration overall) | 39 (Includes patients switched to canakinumab from Week 25 - Week 72)
Completed | 68 | 63
Not Completed | 1 | 3
Not completed — Death | 1 | 1
Not completed — Unsatisfactory therapeutic effect | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Canakinumab 150 mg: Patients received 1 subcutaneous (sc) injection of canakinumab 150 mg and 1 intramuscular (im) injection of placebo to triamcinolone acetonide on Day 1. Patients could receive a re-dose of study drug on demand upon the occurrence of new flares, but re-dosing could not occur until 14 days had elapsed after the previous dose. Patients completing the 12 weeks core study were allowed to continue to be treated in another 12 weeks extension study for any new gout flare on demand with the same treatment as assigned in the core study.
- Triamcinolone Acetonide 40 mg: Patients received 1 intramuscular (im) injection of triamcinolone acetonide 40 mg and 1 subcutaneous (sc) injection of placebo to canakinumab on Day 1. Patients could receive a re-dose of study drug on demand upon the occurrence of new flares, but re-dosing could not occur until 14 days had elapsed after the previous dose. Patients completing the 12 weeks core study were allowed to continue to be treated in another 12 weeks extension study for any new gout flare on demand with the same treatment as assigned in the core study.
- Total: Total of all reporting groups
Arm/Group | Canakinumab 150 mg | Triamcinolone Acetonide 40 mg | Total
Number analyzed (Participants) | 113 | 115 | 228
Age, Continuous [Mean (Standard Deviation); unit: years] — Two patients randomized to canakinumab were not included in the data set (safety set) used to calculate demographic data as they did not receive any study medication and were discontinued from the study on the day of randomization.
  years | 54 (11.18) | 54.6 (10.71) | 54.3 (10.93)
Age, Customized [Number; unit: participants]
  < 65 years | 92 | 92 | 184
  ≥ 65 - 74 years | 16 | 21 | 37
  ≥ 75 years | 5 | 2 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 7 | 19
  Male | 101 | 108 | 209

OUTCOME MEASURES:

1. Primary Outcome: Time to First New Flare
Description: Kaplan-Meier estimates of time to first new flare and confidence intervals were determined. For patients with event, time to event = (date of event - date of first dose of study drug + 1).
  Patients met definition of new flare if they had:
  * Flare in joint, not a previously affected joint (at baseline or during study)
  * Flare in joint previously affected (at baseline or during study) after previous flare in joint has resolved completely.
  Patients did not meet criterion of having new gout flare if:
  · Increasing/renewed gout pain in an affected joint before flare has resolved completely.
Time Frame: 12 weeks
Population: The Full Analysis Set (FAS) consisted of all patients as randomized in the core study who had taken at least one dose of study drug.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Canakinumab 150 mg | Triamcinolone Acetonide 40 mg
Number analyzed (Participants) | 113 | 115
Days | NA [NA to NA] — The median time to first new flare could not be estimated because <50% of patients had a new flare during the time period. | NA [NA to NA] — The median time to first new flare could not be estimated because <50% of patients had a new flare during the time period.

2. Secondary Outcome: Time to at Least a 50% Reduction in Self-assessed Pain Intensity in the Joint Most Affected at Baseline Measured on a Visual Analog Scale (0-100mm VAS)
Description: The Kaplan-Meier estimates of the time to at least a 50% reduction in self-assessed pain intensity in the joint most affected at baseline was determined along with the 95% confidence interval. Patients scored their pain intensity on a 0-100 mm VAS, ranging from no pain (0) to unbearable pain (100). Scores on the 100 mm linear scale were measured to the nearest millimeter from the left. Pain was scored at Baseline; at 6 and 12 hours post-dose; and at 1, 2, 3, 4, 5, 6, and 7 days post-dose.
Time Frame: From baseline to 7 days post dose (randomization)
Population: The Full Analysis Set (FAS) consisted of all patients as randomized in the core study who had taken at least one dose of study drug. Last Observation Carried Forward (LOCF) method was used to impute post dose measurement.
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | Canakinumab 150 mg | Triamcinolone Acetonide 40 mg
Number analyzed (Participants) | 112 | 111
Hours | 48.0 [24.0 to 60.0] | 72.0 [48.0 to 96.0]

3. Secondary Outcome: Time to Complete Resolution of Pain
Description: Patients scored their pain intensity on a 5-point Likert scale (none, mild, moderate, severe, extreme). Complete Resolution of Pain is defined as no pain (None) on the Likert Scale. Pain was scored at Baseline; at 6 and 12 hours post-dose; and at 1, 2, 3, 4, 5, 6, and 7 days post-dose. The Kaplan-Meier estimates of time to complete resolution of self-assessed pain intensity in the joint most affected and their confidence intervals were determined.
Time Frame: 7 days post-dose (randomization)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | Canakinumab 150 mg | Triamcinolone Acetonide 40 mg
Number analyzed (Participants) | 113 | 115
Hours | NA [NA to NA] — The median time to complete resolution could not be estimated because <50% of patients had a complete resolution during the time period. | NA [NA to NA] — The median time to complete resolution could not be estimated because <50% of patients had a complete resolution during the time period.

4. Secondary Outcome: Percentage of Participants With Complete Resolution of Pain
Description: Patients scored their pain intensity on a 5-point Likert scale (none, mild, moderate, severe, extreme). Pain was scored at Baseline; at 6 and 12 hours post-dose; and at 1, 2, 3, 4, 5, 6, and 7 days post-dose. Complete Resolution of Pain is defined as no pain (None) on the Likert Scale. The Kaplan-Meier estimates of cumulative event rate = percentage of participants with event up to the end of the time interval.
Time Frame: 7 days post-dose (randomization)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Canakinumab 150 mg | Triamcinolone Acetonide 40 mg
Number analyzed (Participants) | 113 | 115
Percentage of participants | 34.5 [26.6 to 44.1] | 31.3 [23.7 to 40.6]

5. Secondary Outcome: Percentage of Participants With at Least 1 New Gout Flare During the 12 Weeks
Description: Patients met definition of new flare if they had:
  * Flare in joint, not a previously affected joint (at baseline or during study)
  * Flare in joint previously affected (at baseline or during study) after previous flare in joint has resolved completely.
  Patients did not meet criterion of having new gout flare if:
  · Increasing/renewed gout pain in an affected joint before the flare has resolved completely.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Canakinumab 150 mg | Triamcinolone Acetonide 40 mg
Number analyzed (Participants) | 113 | 115
Percentage of participants | 18.6 | 34.8

6. Secondary Outcome: Mean Number of New Gout Flares Per Patient
Description: as for outcome 5
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: New flares/patient/12 weeks
Arm/Group | Canakinumab 150 mg | Triamcinolone Acetonide 40 mg
Number analyzed (Participants) | 113 | 115
New flares/patient/12 weeks | 0.21 (0.472) | 0.53 (0.892)

7. Secondary Outcome: SF36 Physical Function Score at Week 12
Description: The SF-36 measures the impact of disease on overall quality of life (QoL). This 36-item survey has 8 subscales that can be aggregated into physical- and mental-component summary scores. Scores are standardized with the use of norm-based methods based on an assessment of the general U.S. population free of chronic conditions. Scores range from 1-100 with a mean=50 and a standard deviation=10. A higher score indicates less impact on QoL. A negative change score indicates improvement. An ANCOVA model was used with treatment group and baseline SF-36 physical function subscore as covariates.
Time Frame: Week 12
Population: The Full Analysis Set (FAS) consisted of all patients as randomized in the core study who had taken at least one dose of study drug. Participant observations at Week 12 were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Canakinumab 150 mg | Triamcinolone Acetonide 40 mg
Number analyzed (Participants) | 96 | 92
Units on a scale | 71.76 (2.688) | 71.48 (2.745)

8. Secondary Outcome: Time to First New Flare
Description: Kaplan-Meier (KM) estimates of time to first new flare and confidence intervals were determined. Patients met definition of new flare if they had:
  * Flare in joint, not a previously affected joint (at baseline or during study)
  * Flare in joint previously affected (at baseline or during study) after previous flare in joint has resolved completely.
  Patients did not meet criterion of having new gout flare if:
  · Increasing/renewed gout pain in an affected joint before the flare has resolved completely.
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Canakinumab 150 mg | Triamcinolone Acetonide 40 mg
Number analyzed (Participants) | 113 | 115
Days | NA [NA to NA] — The median time to first new flare could not be estimated because <50% of patients had a new flare during the time period. | 119 [94 to NA] — The upper limit was not estimable in the study as it is longer than the duration of the study (24 weeks).

9. Secondary Outcome: Mean Number of New Gout Flares Per Patient During the 24 Weeks of the Study
Description: as for outcome 5
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: New flares/patient/24 weeks
Arm/Group | Canakinumab 150 mg | Triamcinolone Acetonide 40 mg
Number analyzed (Participants) | 113 | 115
New flares/patient/24 weeks | 0.40 (0.634) | 0.87 (1.104)

10. Secondary Outcome: Time to First Intake of Rescue Medication After the Last Post Baseline Flare.
Description: The Kaplan-Meier estimates of medians and 95% confidence intervals were used to calculate the endpoint.
Time Frame: 72 hours post-dose for the last post-baseline flare (during 24 weeks overall)
Population: The Full Analysis Set (FAS) consisted of all patients as randomized in the core study who had taken at least one dose of study drug. Patients with observations 72 hours post-dose for the last post-baseline flare during 24 weeks were included in analysis.
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | Canakinumab 150 mg | Triamcinolone Acetonide 40 mg
Number analyzed (Participants) | 35 | 43
Hours | NA [12 to NA] — The data were not estimable as <50% patients took rescue medication. | NA [11 to NA] — The data were not estimable as <50% patients took rescue medication.

11. Secondary Outcome: Patient's Assessment of Gout Pain Intensity in the Most Affected Joint on a Visual Analog Scale (VAS) in Extension
Description: Patients scored their pain intensity in the joint most affected at baseline on a 0-100 mm VAS, ranging from no pain (0) to unbearable pain (100). Scores on the 100 mm linear scale were measured to the nearest millimeter from the left. The ANCOVA analysis included treatment group, Baseline VAS score, and body mass index (BMI) at Baseline as covariates.
Time Frame: 72 hours post-dose for the last post-baseline flare (during 24 weeks overall)
Population: The Full Analysis Set (FAS) consisted of all patients as randomized in the core study who had taken at least one dose of study drug. Last Observation Carried Forward (LOCF) method was applied to impute post dose measurements.
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Canakinumab 150 mg | Triamcinolone Acetonide 40 mg
Number analyzed (Participants) | 35 | 41
mm | 34.6 (4.35) | 44.9 (4.01)

12. Secondary Outcome: Percentage of Participants With Maximum Severity of Last Post-baseline Flare (5-point Likert Scale)
Description: Maximum severity is the maximum Likert score recorded after the start of the flare. Participant scored their current pain intensity in the most affected joint of the gout flare on a 5-point Likert Scale (none, mild, moderate, severe, extreme). It participant had a new flare, they also scored the maximum amount of acute gout pain in the most affected joint since the onset of a new flare on 5 point Likert scale (none, mild, moderate, severe, extreme).
Time Frame: Last post-baseline flare (during 24 weeks overall)
Population: The Full Analysis Set (FAS) consisted of all patients as randomized in the core study who had taken at least one dose of study drug. Participants with baseline and last post-baseline observations were included in this analysis.
Measure: Number; unit: Percentage of participants
Arm/Group | Canakinumab 150 mg | Triamcinolone Acetonide 40 mg
Number analyzed (Participants) | 35 | 43
Percentage of participants
  None | 0.0 | 0.0
  Mild | 0.0 | 2.3
  Moderate | 14.3 | 16.3
  Severe | 77.1 | 60.5
  Extreme | 8.6 | 20.9

13. Primary Outcome: Self-assessed Pain Intensity in the Joint Most Affected at Baseline Measured on a Visual Analog Scale (0-100mm VAS)
Description: Patients scored their pain intensity in the joint most affected at baseline on a 0-100 mm VAS, ranging from no pain (0) to unbearable pain (100), at 72 hours post-dose. Scores on the 100 mm linear scale were measured to the nearest millimeter from the left. The ANCOVA analysis included treatment group, Baseline VAS score, and body mass index (BMI) at Baseline as covariates.
Time Frame: 72 hours post-dose (randomization)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Canakinumab 150 mg | Triamcinolone Acetonide 40 mg
Number analyzed (Participants) | 112 | 111
mm | 28.1 (2.42) | 39.5 (2.44)

14. Secondary Outcome: Amount of Rescue Medication Taken
Description: Patients who had difficulty in tolerating their pain were allowed to take rescue medication after the 6-hour post-dose pain assessments as follows:
  * Acetaminophen (paracetamol) 500 mg and/ or codeine 30 mg as required. A maximum of 1 g/dose or 3 g/day of acetaminophen and 30 mg/ dose or 180 mg/day of codeine was allowed.
  * If they had insufficient pain relief, patients were allowed to take a maximum of 30 mg of oral prednisolon as required per day for 2 days followed by up to 20 mg of prednisolone as required subsequent days within 7 days of a gout flare.
Time Frame: 7 days last post-baseline flare (during 24 weeks)
Population: The Full Analysis Set (FAS) consisted of all patients as randomized in the core study who had taken at least one dose of study drug. Patients with observations at 7 days last post-baseline flare were included in this analysis.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Canakinumab 150 mg | Triamcinolone Acetonide 40 mg
Number analyzed (Participants) | 35 | 43
mg
  Acetaminophen | 1931.4 (3266.12) | 2058.1 (3331.33)
  Codeine | 7.7 (25.56) | 46.0 (118.26)
  Prednisolone/Prednisone | 4.1 (17.34) | 21.6 (47.42)

15. Secondary Outcome: Percentage of Participants Who Took Rescue Medication
Description: Patients who had difficulty in tolerating their pain were allowed to take rescue medication after the 6-hour post-dose pain assessments. Permitted rescue medications included acetaminophen 500 mg and/ or codeine 30 mg as needed. If they had insufficient pain relief, patients were allowed to take a maximum of 30 mg of oral prednisolone as needed per day for 2 days followed by up to 20 mg of prednisolone as needed per day for 3 subsequent days within 7 days after randomization or after re-dose/injection administration.
Time Frame: during 12 weeks core, 24 weeks overall
Population: The Full Analysis Set (FAS) consisted of all patients as randomized in core study who had taken at least one dose of study drug. "12 weeks:Core" consisted of patients taking rescue medication during baseline flare of Core study and "24 weeks:Overall" consisted of patients who took rescue medication during last post-baseline flare during 24 weeks.
Measure: Number; unit: Percentage of participants
Arm/Group | Canakinumab 150 mg | Triamcinolone Acetonide 40 mg
Number analyzed (Participants) | 113 | 115
Percentage of participants
  12 weeks :Core (N=113, 115) | 31.0 [NotEst to NotEst] | 52.2 [30 to NotEst]
  24 weeks: Overall (N=35, 43) | 48.6 | 44.2

16. Secondary Outcome: High-sensitivity C-reactive Protein (hsCRP) and Serum Amyloid A Protein (SAA) Levels for Core and 24 Weeks Overall
Description: High sensitivity C-reactive protein (hsCRP) and serum amyloid A (SAA) were determined in blood serum in order to identify the presence of inflammation, to determine its severity, and to monitor the response to treatment. Analytes were measured by a central laboratory. The analysis included treatment group, log-transformed protein level at baseline, and body mass index (BMI) at baseline as covariates.
Time Frame: 72 hours post-dose (randomization), 72 hours post-dose for the last post-baseline flare (during 24 weeks overall)
Population: The Full Analysis Set (FAS) consisted of all patients as randomized in core study who had taken at least one dose of study drug. Patients with baseline flare and data at 72 hours post-dose in core and patients with a new flare and data at 72 hours post-dose for the last post-baseline flare (during 24 weeks overall) were included in this analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/L
Arm/Group | Canakinumab 150 mg | Triamcinolone Acetonide 40 mg
Number analyzed (Participants) | 113 | 115
mg/L
  hsCRP : Core(n= 109, 107) | 4.50 [3.96 to 5.12] | 7.08 [6.22 to 8.07]
  SAA protein : Core (n=105, 106) | 6.77 [5.57 to 8.21] | 17.00 [14.01 to 20.62]
  hsCRP : 24 weeks(n= 31, 32) | 5.18 [3.79 to 7.09] | 7.18 [5.27 to 9.77]
  SAA protein : 24 weeks (n=28, 33) | 11.43 [7.76 to 16.84] | 21.11 [14.78 to 30.16]

17. Secondary Outcome: Physician's Global Assessment of Response to Treatment
Description: The study physician made a global assessment of the patient's response to treatment using a 5-point Likert scale: Very good, good, fair, poor, very poor. The percentage of patients in each category is reported. The physician completed the assessment without viewing any of the patient's assessments (pain intensity [Visual Analog Scale and Likert scale] and patient's global assessment of response to treatment).
Time Frame: 72 hours post-dose (randomization), 72 hours post-dose for the last post-baseline flare (during 24 weeks overall)
Population: The Full Analysis Set (FAS) consisted of all patients as randomized in the core study who had taken at least one dose of study drug. 'N' in each category indicates participants with observations analyzed for this endpoint at specified time points.
Measure: Number; unit: Percentage of participants
Groups:
- Triamcinolone Acetonide 40 mg: Patients received 1 intramuscular (im) injection of triamcinolone acetonide 40 mg and 1 subcutaneous (sc) injection of placebo to canakinumab on Day 1. Patients could receive a re-dose of study drug on demand upon the occurrence of new flares, but re-dosing could not occur until 14 days had elapsed after the previous dose. Patients completing the 12 weeks core study were allowed to continue to be treated in another 12 week extension study for any new gout flare on demand with the same treatment as assigned in the core study.
  Patients under this arm who agreed to continue to 2nd extension period of 12 months, were switched to canakinumab 150 mg sc for any new gout flare during this period
Arm/Group | Canakinumab 150 mg | Triamcinolone Acetonide 40 mg
Number analyzed (Participants) | 113 | 115
Percentage of participants
  Very good (Core) [N=113,110] | 16.8 | 15.5
  Good (Core) [N=113, 110] | 47.8 | 30.0
  Fair (Core) [N= 113, 110] | 26.5 | 32.7
  Poor (Core) [N= 113, 110] | 7.1 | 14.5
  Very poor (Core) [N=113, 110] | 1.8 | 7.3
  Very Good ( 24 weeks) [N=87, 79] | 43.7 | 27.8
  Good (24 weeks) [N=87, 79] | 50.6 | 50.6
  Fair (24 weeks) [N=87, 79] | 5.7 | 17.7
  Poor (24 weeks) [N=87, 79] | 0.0 | 3.8
  Very Poor (24 weeks) [N=87, 79] | 0.0 | 0.0

18. Secondary Outcome: Patient's Global Assessment of Response to Treatment
Description: Patients made a global assessment of response to treatment using a 5-point Likert scale: Excellent, good, acceptable, slight, poor. Percentage of participants in each category for both core and extension periods were measured.
Time Frame: 72 hours post-dose (randomization), 72 hours post-dose for the last post-baseline flare (during 24 weeks overall)
Population: as for outcome 17
Measure: Number; unit: Percentage of participants
Arm/Group | Canakinumab 150 mg | Triamcinolone Acetonide 40 mg
Number analyzed (Participants) | 113 | 115
Percentage of participants
  Excellent (Core) [N=113, 111] | 12.4 | 12.6
  Good (Core) [N=113, 111] | 38.9 | 28.8
  Acceptable (Core) [N=113, 111] | 37.2 | 30.6
  Slight (Core) [N=113, 111] | 8.8 | 12.6
  Poor (Core) [N=113, 111] | 2.7 | 15.3
  Excellent (24 weeks) [N=87, 78] | 31 | 17.9
  Good (24 weeks) [N=87, 78] | 46 | 44.9
  Acceptable (24 weeks) [N=87, 78] | 20.7 | 25.6
  Slight (24 weeks) [N=87, 78] | 1.1 | 9.0
  Poor (24 weeks) [N=87, 78] | 1.1 | 2.6

19. Primary Outcome: Number of Participants With Adverse Events (AE), Death and Serious Adverse Events (24 Weeks Overall)
Description: This was the primary endpoint of both extension studies. Adverse event is defined as any unfavorable and unintended diagnosis, symptom, sign(including an abnormal laboratory finding),syndrome or disease which either occurs during the study, having been absent at baseline, or,if present at baseline, appears to worsen. Serious adverse event is defined as any untoward medical occurrence that results in death, is life threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, or is a congenital anomaly/birth defect.
Time Frame: 24 weeks overall
Population: Safety population consisted of all patients who received study drug in the core study and had at least one post-baseline safety assessment.
Measure: Number; unit: Participants
Groups:
- Triamcinolone Acetonide 40 mg: Patients received 1 intramuscular (im) injection of triamcinolone acetonide 40 mg and 1 subcutaneous (sc) injection of placebo to canakinumab on Day 1. Patients could receive a re-dose of study drug on demand upon the occurrence of new flares, but re-dosing could not occur until 14 days had elapsed after the previous dose. Patients completing the 12 weeks core study were allowed to continue to be treated in another 12 week extension study for any new gout flare on demand with the same treatment as assigned in the core study.
Arm/Group | Canakinumab 150 mg | Triamcinolone Acetonide 40 mg
Number analyzed (Participants) | 113 | 115
Participants
  Adverse Event | 71 | 56
  Death | 0 | 1
  Serious Adverse Event | 11 | 6

20. Secondary Outcome: Physician's Assessment of Tenderness, Swelling, and Erythema of the Most Affected Joint
Description: The study physician assessed the most affected joint for: Tenderness on a 0-3 point scale: No pain, patient states that "there is pain", patient states "there is pain and winces", and patient states "there is pain, winces, and withdraws" on palpation or passive movement of the affected study joint; Swelling on a 0-3 point scale: No swelling, palpable, visible, and bulging beyond the joint margins; and Erythema: Present or absent. The percentage of patients in each category is reported.
Time Frame: 72 hours post-dose (randomization), 72 hours post-dose for the last post-baseline flare (during 24 weeks overall)
Population: as for outcome 17
Measure: Number; unit: Percentage of participants
Arm/Group | Canakinumab 150 mg | Triamcinolone Acetonide 40 mg
Number analyzed (Participants) | 113 | 115
Percentage of participants
  TENDERNESS - No pain (Core) [N=113, 110] | 33.6 | 26.4
  Pain (Core) [N=113, 110] | 56.6 | 51.8
  Pain and winces (Core) [N=113, 110] | 8.0 | 17.3
  Pain,winces,withdraws (Core) [N=113,110] | 1.8 | 4.5
  SWELLING - No swelling (Core) [N=113, 110] | 38.1 | 30.0
  Palpable (Core) [N=113, 110] | 38.9 | 35.5
  Visible (Core) [N=113, 110] | 21.2 | 29.1
  Bulging beyond joint margin (Core) [N=113, 110] | 1.8 | 5.5
  ERYTHEMA - Absent (Core) [N=112, 109] | 78.6 | 65.1
  Present (Core) [N=112, 109] | 21.4 | 34.9
  TENDERNESS - No pain (24 weeks) [N=87, 80] | 82.8 | 85.0
  Pain (24 weeks) [N=87, 80] | 17.2 | 13.8
  Pain and winces (24 weeks) [N=87, 80] | 0.0 | 1.3
  Pain,winces,withdraws (24 weeks) [N=87, 80] | 0.0 | 0.0
  SWELLING - No swelling (24 weeks) [N=87, 80] | 88.5 | 93.8
  Palpable (24 weeks) [N=87, 80] | 8.0 | 5.0
  Visible (24 weeks) [N=87, 80] | 3.4 | 1.3
  Bulging beyond joint margin (24 week)[N=87,80] | 0.0 | 0.0
  ERYTHEMA - Absent (24 weeks) [N=87, 80] | 98.9 | 100
  Present (24 weeks) [N=87, 80] | 1.1 | 0.0

21. Secondary Outcome: Physician's Assessment of Range of Motion of the Most Affected Joint
Description: The study physician assessed the range of motion of the most affected joint for range of motion on a 5-point Likert scale: Normal, mildly restricted, moderately restricted, severely restricted, immobilized. The percentage of patients in each category is reported.
Time Frame: 72 hours post-dose (randomization), 72 hours post-dose for the last post-baseline flare (24 weeks overall)
Population: Full Analysis Set (FAS): All patients that received study drug. 'N' in each category indicates participants with observations analyzed for this endpoint at specified time points.
Measure: Number; unit: Percentage of participants
Arm/Group | Canakinumab 150 mg | Triamcinolone Acetonide 40 mg
Number analyzed (Participants) | 113 | 115
Percentage of participants
  Normal (Core) [N=113, 111] | 25.7 | 31.5
  Mildly restricted (Core) [N=113, 111] | 50.4 | 29.7
  Moderately restricted (Core) [N=113, 111] | 21.2 | 27.0
  Severely restricted (Core) [N=113, 111] | 2.7 | 8.1
  Immobilized (Core) [N=113, 111] | 0.0 | 3.6
  Normal (24 weeks) [N=87, 79] | 66.7 | 65.8
  Mildly restricted (24 weeks) [N=87, 79] | 31.0 | 29.1
  Moderately Restricted (24 weeks) [N=87, 79] | 2.3 | 3.8
  Severely Restricted (24 weeks) [N=87, 79] | 0.0 | 1.3
  Immobilized (24 weeks) [N=87, 79] | 0.0 | 0.0

22. Secondary Outcome: Patient's Assessment of Gout Pain Intensity in the Most Affected Joint (Likert Scale)
Description: Participant scored their current pain intensity in the most affected joint of the gout flare on a 5-point Likert Scale (none, mild, moderate, severe, extreme). It participant had a new flare, they also scored the maximum amount of acute gout pain in the most affected joint since the onset of a new flare on 5 point Likert scale (none, mild, moderate, severe, extreme).
Time Frame: 7 days post dose (randomization), 24 weeks post-dose
Population: Full Analysis Set includes all patients that received study drug. 'N' in each category indicates participants with observations analyzed for this endpoint at specified time points.
Measure: Number; unit: Percentage of participants
Arm/Group | Canakinumab 150 mg | Triamcinolone Acetonide 40 mg
Number analyzed (Participants) | 113 | 115
Percentage of participants
  None (7 days post-dose) [N= 110, 107] | 32.7 | 28.0
  Mild (7 days post-dose) [N= 110, 107] | 48.2 | 41.1
  Moderate (7 days post-dose) [N= 110, 107] | 16.4 | 16.8
  Severe (7 days post-dose) [N= 110, 107] | 2.7 | 12.1
  Extreme (7 days post-dose) [N= 110, 107] | 0.0 | 1.9
  None (24 weeks post-dose) [N= 85, 78] | 47.1 | 46.2
  Mild (24 weeks post-dose) [N= 85, 78] | 38.8 | 37.2
  Moderate (24 weeks post-dose) [N= 85, 78] | 12.9 | 15.4
  Severe (24 weeks post-dose) [N= 85, 78] | 1.2 | 1.3
  Extreme (24 weeks post-dose) [N= 85, 78] | 0.0 | 0.0

23. Secondary Outcome: Time to First New Flare: Survival Analysis by Treatment (72 Weeks Overall)
Description: as for outcome 1
Time Frame: 72 weeks overall
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Groups:
- Triamcinolone Acetonide 40 mg: Patients received 1 intramuscular (im) injection of triamcinolone acetonide 40 mg and 1 subcutaneous (sc) injection of placebo to canakinumab on Day 1. Patients could receive a re-dose of study drug on demand upon the occurrence of new flares, but re-dosing could not occur until 14 days had elapsed after the previous dose. Patients completing the 12 weeks core study were allowed to continue to be treated in another 12 weeks extension study for any new gout flare on demand with the same treatment as assigned in the core study. Patients under this arm who agreed to continue to 2nd extension period of 12 months, were switched to canakinumab 150 mg sc for any new gout flare during this period
Arm/Group | Canakinumab 150 mg | Triamcinolone Acetonide 40 mg
Number analyzed (Participants) | 113 | 115
days | 222.0 [190.0 to 274.0] | 119.0 [94 to 224.0]

24. Secondary Outcome: Flare Rate Per Year
Description: Flare rate was calculated as the number of new flares over the period of observation in years. Flare rate was calculated using only those new flares before switching to canakinumab.
  Patients met definition of new flare if they had:
  * Flare in joint, not a previously affected joint (at baseline or during study)
  * Flare in joint previously affected (at baseline or during study) after previous flare in joint has resolved completely.
  Patients did not meet criterion of having new gout flare if:
  · Increasing/renewed gout pain in an affected joint before the flare has resolved completely.
Time Frame: 72 weeks overall
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: New flares per patient per year
Groups:
- Triamcinolone Acetonide 40 mg: Patients received 1 intramuscular (im) injection of triamcinolone acetonide 40 mg and 1 subcutaneous (sc) injection of placebo to canakinumab on Day 1. Patients could receive a re-dose of study drug on demand upon the occurrence of new flares, but re-dosing could not occur until 14 days had elapsed after the previous dose. Patients completing the 12 weeks core study were allowed to continue to be treated in another 12 week extension study for any new gout flare on demand with the same treatment as assigned in the core study.
  Patients under this arm who agreed to continue to 2nd extension period of 12 months, were switched to canakinumab 150 mg sc for any new gout flare during this period. Note that flare rate was calculated using only those new flares before switching.
Arm/Group | Canakinumab 150 mg | Triamcinolone Acetonide 40 mg
Number analyzed (Participants) | 113 | 115
New flares per patient per year | 1.16 (1.511) [0.97 to 1.51] | 2.81 (4.399) [1.72 to 2.71]

25. Secondary Outcome: High-sensitivity C-reactive Protein (hsCRP) Levels for Patients Re-treated With or Switched to Canakinumab
Description: High sensitivity C-reactive protein (hsCRP) levels were determined in blood serum in order to identify the presence of inflammation, to determine its severity, and to monitor the response to treatment. Analytes were measured by a central laboratory. The treatment effect reported for canakinumab arm was for last post-baseline flare after re-treated with canakinumab and for patient which switched to Canakinumab arm was for first post-baseline flare after receiving the first dose of canakinumab.
Time Frame: 24 hours, 72 hours, 7 days, 4 weeks, 8 weeks and 12 weeks post-dose for the last post-baseline flare for patients re-treated with canakinumab or first post-baseline flare treated with canakinumab for patients switched treatment (during 72 weeks overall)
Population: Modified Analysis Set (MAS) consists of all FAS patients who were either re-treated or switched to canakinumab during 72 weeks. At each timepoint only patients with a value at both baseline flare and the new flare are included
Measure: Mean (Standard Deviation); unit: mg/L
Groups:
- Randomized to Canakinumab and Re-treated With Canakinumab: Patients received 1 subcutaneous (sc) injection of canakinumab 150 mg and 1 intramuscular (im) injection of placebo to triamcinolone acetonide on Day 1. Patients could receive a re-dose of study drug on demand upon the occurrence of new flares, but re-dosing could not occur until 14 days had elapsed after the previous dose. Patients completing the 12 weeks core study were allowed to continue to be treated in another 12 weeks extension study for any new gout flare on demand with the same treatment as assigned in the core study.
- Randomized to Triamcinolone and Switched to Canakinumab: Patients received 1 intramuscular (im) injection of triamcinolone acetonide 40 mg and 1 subcutaneous (sc) injection of placebo to canakinumab on Day 1. Patients could receive a re-dose of study drug on demand upon the occurrence of new flares, but re-dosing could not occur until 14 days had elapsed after the previous dose. Patients completing the 12 weeks core study were allowed to continue to be treated in another 12 week extension study for any new gout flare on demand with the same treatment as assigned in the core study.
  Patients under this arm who agreed to continue to 2nd extension period of 12 months, were switched to canakinumab 150 mg sc for any new gout flare during this period
Arm/Group | Randomized to Canakinumab and Re-treated With Canakinumab | Randomized to Triamcinolone and Switched to Canakinumab
Number analyzed (Participants) | 69 | 39
mg/L
  24 hours post dose (n= 45, 24) | 28.9 (42.26) | 26.0 (29.07)
  72 hours post dose (n=45, 34) | 10.6 (14.69) | 7.0 (8.06)
  7 days post dose (n=67, 39) | 3.3 (3.38) | 3.2 (3.57)
  4 weeks post dose (n=52, 35) | 9.2 (48.57) | 3.2 (4.95)
  8 weeks post dose (n=45, 37) | 2.6 (3.00) | 3.0 (6.74)
  12 weeks post dose (n=42, 33) | 6.5 (12.99) | 4.3 (11.90)

26. Secondary Outcome: Serum Amyloid A Protein (SAA) Levels for Patients Re-treated With or Switched to Canakinumab
Description: Serum Amyloid A Protein (SAA) levels were determined in blood serum in order to identify the presence of inflammation, to determine its severity, and to monitor the response to treatment. Analytes were measured by a central laboratory. The treatment effect reported for canakinumab arm was for last post-baseline flare after re-treated with canakinumab and for patient which switched to Canakinumab arm was for first post-baseline flare after receiving the first dose of canakinumab.
Time Frame: as for outcome 25
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Randomized to Canakinumab and Re-treated With Canakinumab | Randomized to Triamcinolone and Switched to Canakinumab
Number analyzed (Participants) | 69 | 39
mg/L
  24 hours post dose (n= 45, 27) | 151.4 (310.09) | 86.5 (188.46)
  72 hours post dose (n=45, 36) | 42.5 (116.89) | 26.9 (73.37)
  7 days post dose (n=67, 39) | 5.4 (8.83) | 4.9 (6.56)
  4 weeks post dose (n=52, 35) | 31.0 (193.64) | 8.5 (19.75)
  8 weeks post dose (n=45, 37) | 4.2 (4.26) | 5.4 (8.36)
  12 weeks post dose (n=42, 33) | 10.7 (24.62) | 7.8 (22.98)

27. Primary Outcome: Number of Participants With Adverse Events (AE), Death and Serious Adverse Events (72 Weeks Overall)
Description: as for outcome 19
Time Frame: 72 weeks overall
Population: as for outcome 19
Measure: Number; unit: Participants
Groups:
- All Randomized to Canakinumab: Patients received 1 subcutaneous (sc) injection of canakinumab 150 mg and 1 intramuscular (im) injection of placebo to triamcinolone acetonide on Day 1. Patients could receive a re-dose of study drug on demand upon the occurrence of new flares, but re-dosing could not occur until 14 days had elapsed after the previous dose. Patients completing the 12 weeks core study were allowed to continue to be treated in another 12 weeks extension study for any new gout flare on demand with the same treatment as assigned in the core study.
  After completing the first extension study, patients were offered to enter the second extension study, whereby all patients were treated open-label "on demand" with canakinumab 150 mg sc upon new flare for 1 year for a total duration of 18 months following randomization in the core study.
- Randomized to Canakinumab :Before Re-treated With Canakinumab: All patients who were randomized to Canakinumab in core study period received 1 subcutaneous (sc) injection of canakinumab 150 mg and 1 intramuscular (im) injection of placebo to triamcinolone acetonide on Day 1 but experienced adverse events before re-treated with canakinumab
- Randomized to Canakinumab :After Re-treated With Canakinumab: All patients who were randomized to Canakinumab in core study period received 1 subcutaneous (sc) injection of canakinumab 150 mg and 1 intramuscular (im) injection of placebo to triamcinolone acetonide on Day 1 but experienced adverse events after re-treated with canakinumab
- Randomized to Triamcinolone Acetonide (Triam): Patients received 1 intramuscular (im) injection of triamcinolone acetonide 40 mg and 1 subcutaneous (sc) injection of placebo to canakinumab on Day 1. Patients could receive a re-dose of study drug on demand upon the occurrence of new flares, but re-dosing could not occur until 14 days had elapsed after the previous dose. Patients completing the 12 weeks core study were allowed to continue to be treated in another 12 week extension study for any new gout flare on demand with the same treatment as assigned in the core study.
  Patients under this arm who agreed to continue to 2nd extension period of 12 months, were switched to canakinumab 150 mg sc for any new gout flare during this period. AE/SAE were only assigned to this group before being switched to canakinumab
- Randomized to Triam: Before Switched to Canakinumab: All patients who were randomized to triamcinolone acetonide (Triam) received 1 intramuscular (im) injection of triamcinolone acetonide 40 mg and 1 subcutaneous (sc) injection of placebo to canakinumab on Day 1, experienced adverse event before switched to canakinumab
- Randomized to Triam: After Switched to Canakinumab: All patients who were randomized to triamcinolone acetonide (Triam) received 1 intramuscular (im) injection of triamcinolone acetonide 40 mg and 1 subcutaneous (sc) injection of placebo to canakinumab on Day 1, experienced adverse event after switched to canakinumab
Arm/Group | All Randomized to Canakinumab | Randomized to Canakinumab :Before Re-treated With Canakinumab | Randomized to Canakinumab :After Re-treated With Canakinumab | Randomized to Triamcinolone Acetonide (Triam) | Randomized to Triam: Before Switched to Canakinumab | Randomized to Triam: After Switched to Canakinumab
Number analyzed (Participants) | 113 | 69 | 69 | 115 | 39 | 39
Participants
  Adverse Event | 76 | 41 | 38 | 60 | 20 | 19
  Death | 1 | 0 | 1 | 2 | 0 | 0
  Serious Adverse Event | 19 | 6 | 8 | 11 | 2 | 0

28. Secondary Outcome: Physician's Global Assessment of Response to Treatment for Patients Re-treated or Switched to Canakinumab
Description: The study physician made a global assessment of the patient's response to treatment using a 5-point Likert scale: Very good, good, fair, poor, very poor. The percentage of patients in each category is reported. The physician completed the assessment without viewing any of the patient's assessments (pain intensity [Visual Analog Scale and Likert scale] and patient's global assessment of response to treatment). The treatment effect reported for canakinumab arm was for last post-baseline flare after re-treated with canakinumab and for patient which switched to Canakinumab arm was for first post-baseline flare after receiving the first dose of canakinumab.
Time Frame: 72 hours post-dose , 7 days post-dose for the last post-baseline flare for patients re-treated with canakinumab or first post-baseline flare treated with canakinumab for patients switched treatment (during 72 weeks overall)
Population: as for outcome 25
Measure: Number; unit: Percentage of participants
Groups:
- Randomized to Canakinumab and Re-treated With Canakinumab: Patients received 1 subcutaneous (sc) injection of canakinumab 150 mg and 1 intramuscular (im) injection of placebo to triamcinolone acetonide on Day 1. Patients could receive a re-dose of study drug on demand upon the occurrence of new flares, but re-dosing could not occur until 14 days had elapsed after the previous dose. Patients completing the 12 weeks core study were allowed to continue to be treated in another 12 weeks extension study for any new gout flare on demand with the same treatment as assigned in the core study.
  After completing the first extension study, patients were offered to enter the second extension study, whereby all patients were treated open-label "on demand" with canakinumab 150 mg sc upon new flare for 1 year for a total duration of 18 months following randomization in the core study.
Arm/Group | Randomized to Canakinumab and Re-treated With Canakinumab | Randomized to Triamcinolone and Switched to Canakinumab
Number analyzed (Participants) | 69 | 39
Percentage of participants
  Very good (72 hours post dose) (n=61, 34) | 21.3 | 22.9
  Good (72 hours post dose) (n=61, 34) | 41.0 | 57.1
  Fair (72 hours post dose) (n=61, 34) | 31.1 | 17.1
  Poor (72 hours post dose) (n=61, 34) | 6.6 | 2.9
  Very poor (72 hours post dose) (n=61, 34) | 0.0 | 0.0
  Very Good (7 days post dose) (n=68, 34) | 36.8 | 33.3
  Good (7 days post dose) (n=68, 34) | 52.9 | 63.9
  Fair (7 days post dose) (n=68, 34) | 10.3 | 0.0
  Poor (7 days post dose) (n=68, 34) | 0.0 | 0.0
  Very Poor (7 days post dose) (n=68, 34) | 0.0 | 2.8

29. Secondary Outcome: Patient's Assessment of Gout Pain Intensity in the Currently Most-affected Joint (Likert Scale)
Description: Participant scored their current pain intensity in the most affected joint of the gout flare on a 5-point Likert Scale (none, mild, moderate, severe, extreme). It participant had a new flare, they also scored the maximum amount of acute gout pain in the most affected joint since the onset of a new flare on 5 point Likert scale (none, mild, moderate, severe, extreme). The treatment effect reported for canakinumab arm was for last post-baseline flare after re-treated with canakinumab and for patient which switched to Canakinumab arm was for first post-baseline flare after receiving the first dose of canakinumab.
Time Frame: 72 hours post-dose , 7 days post dose for the last post-baseline flare for patients re-treated with canakinumab or the first post-baseline flare treated with canakinumab for patients who switched treatment (during 72 weeks overall)
Population: as for outcome 25
Measure: Number; unit: Percentage of participants
Arm/Group | Randomized to Canakinumab and Re-treated With Canakinumab | Randomized to Triamcinolone and Switched to Canakinumab
Number analyzed (Participants) | 69 | 39
Percentage of participants
  None (72 hours post dose) (n=66, 39) | 19.7 | 20.5
  Mild (72 hours post dose) (n=66, 39) | 30.0 | 61.5
  Moderate (72 hours post dose) (n=66, 39) | 45.5 | 15.4
  Severe (72 hours post dose) (n=66, 39) | 4.5 | 0.0
  Extreme (72 hours post dose) (n=66, 39) | 0.0 | 2.6
  None (7 days post dose) (n=65, 35) | 41.5 | 57.1
  Mild (7 days post dose) (n=65, 35) | 38.5 | 34.3
  Moderate (7 days post dose) (n=65, 35) | 18.5 | 5.7
  Severe (7 days post dose) (n=65, 35) | 1.5 | 0.0
  Extreme (7 days post dose) (n=65, 35) | 0.0 | 2.9

30. Secondary Outcome: Patient's Global Assessment of Response to Treatment for Patients Re-treated or Switched to Canakinumab
Description: Patients made a global assessment of response to treatment using a 5-point Likert scale: Excellent, good, acceptable, slight, poor. Percentage of participants in each category for both core and extension periods were measured. The treatment effect reported for canakinumab arm was for last post-baseline flare after re-treated with canakinumab and for patient which switched to Canakinumab arm was for first post-baseline flare after receiving the first dose of canakinumab.
Time Frame: as for outcome 29
Population: as for outcome 25
Measure: Number; unit: Percentage of participants
Arm/Group | Randomized to Canakinumab and Re-treated With Canakinumab | Randomized to Triamcinolone and Switched to Canakinumab
Number analyzed (Participants) | 69 | 39
Percentage of participants
  Excellent (72 hours post dose) (n=60, 36) | 15.0 | 19.4
  Good (72 hours post dose) (n=60, 36) | 26.7 | 44.4
  Acceptable (72 hours post dose) (n=60, 36) | 50.0 | 27.8
  Slight (72 hours post dose) (n=60, 36) | 6.7 | 2.8
  Poor (72 hours post dose) (n=60, 36) | 1.7 | 5.6
  Excellent (7 days post dose) (n=68, 36) | 23.5 | 27.8
  Good (7 days post dose) (n=68, 36) | 41.2 | 52.8
  Acceptable (7 days post dose) (n=68, 36) | 27.9 | 16.7
  Slight (7 days post dose) (n=68, 36) | 7.4 | 2.8
  Poor (7 days post dose) (n=68, 36) | 0.0 | 0.0

31. Secondary Outcome: Physician's Assessment of Joint Tenderness for Patients Re-treated or Switched to Canakinumab
Description: The study physician assessed the most affected joint for: Tenderness on a 0-3 point scale: No pain, patient states that "there is pain", patient states "there is pain and winces", and patient states "there is pain, winces, and withdraws" on palpation or passive movement of the affected study joint; The percentage of patients in each category is reported. The treatment effect reported for canakinumab arm was for last post-baseline flare after re-treated with canakinumab and for patient which switched to Canakinumab arm was for first post-baseline flare after receiving the first dose of canakinumab.
Time Frame: 72 hours post-dose , 7 days post dose last post-baseline flare for patients re-treated with canakinumab or the first post-baseline flare treated with canakinumab for patients who switched treatment (during 72 weeks overall)
Population: as for outcome 25
Measure: Number; unit: Percentage of participants
Arm/Group | Randomized to Canakinumab and Re-treated With Canakinumab | Randomized to Triamcinolone and Switched to Canakinumab
Number analyzed (Participants) | 69 | 39
Percentage of participants
  No Pain (72 hours post dose) (n=61, 35) | 27.9 | 28.6
  Pain (72 hours post dose) (n=61, 35) | 54.1 | 68.6
  Pain and winces (72 hours post dose) (n=61, 35) | 16.4 | 2.9
  Pain, winces, withdraw(72 hrs post dose)(n=61, 35) | 1.6 | 0.0
  No pain (7 days post dose) (n=68, 36) | 52.9 | 69.4
  Pain (7 days post dose) (n=68, 36) | 44.1 | 27.8
  Pain and winces (7 days post dose) (n=68, 36) | 2.9 | 2.8
  Pain, winces, withdraw(72 hrs post dose)(n=61, 36) | 0.0 | 0.0

32. Secondary Outcome: Physician's Assessment of Joint Swelling for Patients Re-treated or Switched to Canakinumab
Description: The study physician assessed the most affected joint for: Swelling on a 0-3 point scale: No swelling, palpable, visible, and bulging beyond the joint margins; The percentage of patients in each category is reported. The treatment effect reported for canakinumab arm was for last post-baseline flare after re-treated with canakinumab and for patient which switched to Canakinumab arm was for first post-baseline flare after receiving the first dose of canakinumab.
Time Frame: as for outcome 31
Population: as for outcome 25
Measure: Number; unit: Percentage of participants
Arm/Group | Randomized to Canakinumab and Re-treated With Canakinumab | Randomized to Triamcinolone and Switched to Canakinumab
Number analyzed (Participants) | 69 | 39
Percentage of participants
  No Pain (72 hours post dose) (n=61, 35) | 29.5 | 42.9
  Pain (72 hours post dose) (n=61, 35) | 42.6 | 48.6
  Pain and winces (72 hours post dose) (n=61, 35) | 24.6 | 8.6
  Pain, winces, withdraw(72 hrs post dose)(n=61, 35) | 3.3 | 0.0
  No pain (7 days post dose) (n=68, 36) | 64.7 | 75.0
  Pain (7 days post dose) (n=68, 36) | 25.0 | 16.7
  Pain and winces (7 days post dose) (n=68, 36) | 7.4 | 5.6
  Pain, winces, withdraw(72 hrs post dose)(n=68, 36) | 2.9 | 2.8

33. Secondary Outcome: Physician's Assessment of Erythema for Patients Re-treated or Switched to Canakinumab
Description: The study physician assessed the most affected joint for Erythema: Present or absent. The percentage of patients in each category is reported. The treatment effect reported for canakinumab arm was for last post-baseline flare after re-treated with canakinumab and for patient which switched to Canakinumab arm was for first post-baseline flare after receiving the first dose of canakinumab.
Time Frame: as for outcome 29
Population: as for outcome 25
Measure: Number; unit: Percentage of participants
Arm/Group | Randomized to Canakinumab and Re-treated With Canakinumab | Randomized to Triamcinolone and Switched to Canakinumab
Number analyzed (Participants) | 69 | 39
Percentage of participants
  Absent (72 hours post dose) (n=61, 35) | 82.0 | 80.0
  Present (72 hours post dose) (n=61, 35) | 18.0 | 20.0
  Absent (7 days post dose) (n=67, 36) | 95.5 | 94.4
  Present (7 days post dose) (n=67, 36) | 4.5 | 5.6

ADVERSE EVENTS:
Groups:
- All Randomized to Triamcinolone Acetonide (Triam): Patients received 1 intramuscular (im) injection of triamcinolone acetonide 40 mg and 1 subcutaneous (sc) injection of placebo to canakinumab on Day 1. Patients could receive a re-dose of study drug on demand upon the occurrence of new flares, but re-dosing could not occur until 14 days had elapsed after the previous dose. Patients completing the 12 weeks core study were allowed to continue to be treated in another 12 week extension study for any new gout flare on demand with the same treatment as assigned in the core study.
  Patients under this arm who agreed to continue to 2nd extension period of 12 months, were switched to canakinumab 150 mg sc for any new gout flare during this period. AE/SAE were only assigned to this group before being switched to canakinumab
Arm/Group | All Randomized to Canakinumab | Randomized to Canakinumab :Before Re-treated With Canakinumab | Randomized to Canakinumab :After Re-treated With Canakinumab | All Randomized to Triamcinolone Acetonide (Triam) | Randomized to Triam: Before Switched to Canakinumab | Randomized to Triam: After Switched to Canakinumab
Serious Adverse Events (participants affected / at risk) | 19/113 | 6/69 | 8/69 | 11/115 | 2/39 | 0/39
Other Adverse Events (participants affected / at risk) | 47/113 | 19/69 | 19/69 | 22/115 | 7/39 | 12/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Randomized to Canakinumab (N=113) | Randomized to Canakinumab :Before Re-treated With Canakinumab (N=69) | Randomized to Canakinumab :After Re-treated With Canakinumab (N=69) | All Randomized to Triamcinolone Acetonide (Triam) (N=115) | Randomized to Triam: Before Switched to Canakinumab (N=39) | Randomized to Triam: After Switched to Canakinumab (N=39)
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 1 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Angina unstable (Cardiac disorders) | 1 | 0 | 1 | 1 | 0 | 0
Arrhythmia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 1 | 0 | 0 | 0 | 0
Glaucoma (Eye disorders) | 1 | 1 | 0 | 0 | 0 | 0
Retinal artery occlusion (Eye disorders) | 1 | 1 | 0 | 0 | 0 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Periproctitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Device dislocation (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Abscess jaw (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Endocarditis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Pneumococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 1 | 0 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Meniscus lesion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Prostatic specific antigen increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 0 | 2 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0
Radiculopathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Spinal cord ischaemia (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0
Vertebrobasilar insufficiency (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 0 | 0
Renal colic (Renal and urinary disorders) | 1 | 0 | 1 | 1 | 0 | 0
Renal failure chronic (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Renal impairment (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Randomized to Canakinumab (N=113) | Randomized to Canakinumab :Before Re-treated With Canakinumab (N=69) | Randomized to Canakinumab :After Re-treated With Canakinumab (N=69) | All Randomized to Triamcinolone Acetonide (Triam) (N=115) | Randomized to Triam: Before Switched to Canakinumab (N=39) | Randomized to Triam: After Switched to Canakinumab (N=39)
Bronchitis (Infections and infestations) | 3 | 1 | 1 | 4 | 3 | 3
Influenza (Infections and infestations) | 5 | 1 | 4 | 1 | 0 | 1
Nasopharyngitis (Infections and infestations) | 8 | 4 | 2 | 2 | 1 | 2
Upper respiratory tract infection (Infections and infestations) | 3 | 2 | 1 | 3 | 2 | 1
Gamma-glutamyltransferase increased (Investigations) | 6 | 3 | 1 | 4 | 1 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 2
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 5 | 4 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 2 | 5 | 2 | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 4 | 2 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 7 | 1 | 2 | 2 | 0 | 0
Headache (Nervous system disorders) | 8 | 3 | 2 | 2 | 0 | 1
Hypertension (Vascular disorders) | 13 | 5 | 7 | 10 | 3 | 3

LIMITATIONS AND CAVEATS:
Bioanalytical results: With analytical method used, anti-canakinumab antibodies were detected in 10 patients. However, no patients showed any unexpected PK/ PD profile nor had adverse events suggestive of immunogenicity.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.